CLINICAL TRIAL: NCT05216978
Title: Proof-of-Concept Trial of a Positive Psychology Intervention for Caregivers of Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Proof-of-Concept Trial of a Positive Psychology Intervention for Caregivers of Patients Undergoing HSCT
Acronym: PATH-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Hermioni L.Amonoo, MD, MPP, MPH, Director, Well-Being and Cancer Research Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-596
Record Dates: First submitted 2021-12-20; First posted 2022-02-01 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Caregiver; Hematologic Malignancy
Keywords: Positive Psychology Intervention; Hematopoietic Stem Cell Transplant; Caregivers of Patients with Cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants will receive the PATH intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PATH Intervention (Experimental): Participants in the PATH Intervention arm will receive psychosocial support phone calls during week 1 through 9 following enrollment.
  After consent procedures, participants will begin an 9-week positive-psychology program involving weekly calls with an interventionist and exercises (i.e. writing a letter of gratitude, identifying personal strengths, planning meaningful and enjoyable activities).
  Self-assessment questionnaires to measure positive affect, health behaviors, and overall function before and after completing the Positive Psychology Intervention.
  Interventions: Behavioral: Positive Psychology Intervention

INTERVENTIONS:
Behavioral: Positive Psychology Intervention — Weekly phone calls with the study interventionist and positive psychology exercises over an 9-week period. The positive psychology program exercises include three modules: gratitude-based activities, strength-based activities, and meaning-based activities.

SUMMARY:
Caregivers (i.e., family and friends) of patients with cancer are essential in providing care during cancer treatment. For patients who are undergoing a hematopoietic stem cell transplant/transplantation (HSCT) as treatment for their cancer, caregivers are even more crucial before, during, and after their transplantation. Although HSCT is potentially curative for some patients with blood cancers, the treatment is intensive and accompanied by a prolonged hospitalization as patients recover from the toxic side-effects of chemotherapy and medical complications from the transplantation. Unsurprisingly, during the entire transplantation process, caregiver burden is high as caregivers witness and support their loved ones through multiple treatment-related complications, management of ongoing physical symptoms, and complex medication schedules. Caregiver burden leads to poor health outcomes including poor caregiver quality of life, fatigue, depression, anxiety, impaired physical health, and low levels of resilience and positive emotions. Reducing distress and enhancing positive emotions can both reduce caregiver burden and improve caregiver quality of life. However, the few interventions in the HSCT caregiver population have mostly focused on mitigating distress, despite strong evidence that enhancing positive emotions in caregivers reduces caregiver burden and promotes physical and psychological health. To address this gap, we hope to develop and test an intervention that emphasizes positive emotions in caregivers of HSCT recipients. A scalable and accessible positive emotion-based intervention tailored to the unique needs of HSCT recipients' caregivers provides a new line of behavioral intervention resources that could offer benefit to both caregivers and patients and could be generalizable to other cancer caregivers.

DETAILED DESCRIPTION:
The proposed project (PATH-C) entails two phases:

1. Phase one is an open-pilot trial in 5 caregivers of patients undergoing HSCT to refine the PATH intervention.
2. Phase two is single-arm open-pilot trial evaluating the feasibility and acceptability of the PATH intervention in 20 caregivers of patients undergoing HSCT.

All participants will be approached in-person at the routine HSCT patient consent clinic visit or, with patient permission, over the phone if the caregiver is not physically present at the consent visit for eligibility determination. Interested participants will be screened based on the inclusion/exclusion criteria and verbal consent will be obtained.

Upon consent to participate in the study, participants in both phases will be asked to complete baseline questionnaires either in-person, over the phone, or via a REDCap survey link to participants. After baseline assessments are completed, participants will be given an intervention manual with 9-weekly positive psychology (PP) exercises and an explanation of the exercises and intervention.

All participants in Phases 1 and 2 will be asked to complete the 9-weekly PP exercises starting after the baseline questionnaires (i.e., after the patient transplant consent visit) are completed in the pre-transplant phase and to speak with the study interventionist, a trained clinical research coordinator (CRC), weekly. Immediately after the completion of each exercise, participants will rate the ease of exercise completion, overall utility of the exercise, and their current levels of positive affect. After the Week 9 intervention phone session, all participants in both phases will complete another set of self-assessment questionnaires either over the phone, in-person at a routine clinic visit, or via a REDCap survey link emailed to participants. Additionally, participants will be asked to complete a recorded exit interview over the phone. These individual, semi-structured exit interviews will elicit feedback about the intervention (e.g., relevance and applicability of the chosen PP exercises, intervention length, timing, and delivery), study procedures, and questionnaires. Exit interviews will be recorded, transcribed, coded and thematically analyzed. At study completion, we will inquire about participants' potential interest in being contacted about our future studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregivers (≥18 years) of patients undergoing allogeneic hematopoietic stem cell transplant (HSCT) at Dana-Farber Cancer Institute (DCFI).
* A relative or a friend who either lives with the patient or has in-person contact with him or her at least twice per week and is identified as the primary caregiver for HSCT.
* Ability to speak English and able to complete questionnaires with minimum assistance of an interpreter.

Exclusion Criteria:

* Cognitive deficits impeding a caregiver's ability to provide informed consent or participate adequately in the study assessed via a commonly used 6-item cognitive assessment, the Brief Interview for Mental Status (BIMS) screening tool, which is sensitive and specific for screening for cognitive impairment in research subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermioni L Amonoo, MD, MPP, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber/Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor, Investigator, or designee. The protocol and statistical analysis plan will be made available on ClinicalTrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the study investigator at hermioni_amonoo@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although the study was divided into two phases under a single open-arm study, participants in both phases received the same study procedures so data reported represents patients in both two phases. Considering this is an open-pilot study, we recruited continuously for the study without distinguishing phases. All participants received the positive psychology intervention.
Groups:
- PATH Intervention: Participants in the PATH Intervention arm will receive psychosocial support phone calls during week 1 through 9 following enrollment.
  After consent procedures, participants will begin an 9-week positive-psychology program involving weekly calls with an interventionist and exercises (i.e. writing a letter of gratitude, identifying personal strengths, planning meaningful and enjoyable activities).
  Self-assessment questionnaires to measure positive affect, health behaviors, and overall function before and after completing the Positive Psychology Intervention.
  Positive Psychology Intervention: Weekly phone calls with the study interventionist and positive psychology exercises over an 9-week period. The positive psychology program exercises include three modules: gratitude-based activities, strength-based activities, and meaning-based activities.
Period: Overall Study
Arm/Group | PATH Intervention
Started | 23
Completed | 15
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Baseline data is reported for participants who completed follow-up measures and exit interviews
Arm/Group | PATH Intervention
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Relationship Status [Count of Participants; unit: Participants]
  Married/living together | 12
  Single | 1
  Separated/divorced | 1
  Missing | 1
Religion [Count of Participants; unit: Participants]
  Agnostic | 3
  Catholic Christian | 6
  Other Christian | 3
  Jewish | 1
  None | 1
  Missing | 1
Education [Count of Participants; unit: Participants]
  High school diploma | 2
  Some college | 2
  College degree | 6
  Some postgraduate/professional education | 2
  Postgraduate/professional degree | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the PATH Intervention
Description: Feasibility of the refined PATH intervention and our assessment battery in caregivers of patients who have undergone hematopoietic stem cell transplant (HSCT) using a single-arm trial.
Time Frame: 9 weeks
Population: The analysis populations are as follows.
  Feasibility:
  Enrollment - 49 eligible participants were approached and 23 participants were enrolled. Of the 23 participants who enrolled. 8 participants did not start PATH: 3 withdrew from the study and 5 were lost to follow-up. For the feasibility analysis, the analysis population denominator is 15 participants who started PATH.
Measure: Number; unit: participants
Arm/Group | PATH Intervention
Number analyzed (Participants) | 15
participants
  Number of participants who completed at least 6/9 intervention sessions | 15
  Number of participants who completed all 9/9 intervention sessions | 13
  Number of participants who completed baseline and follow-up assessment battery | 15

2. Primary Outcome: Acceptability Rate
Description: At the end of each weekly intervention session, acceptability was measured with ratings of ease and utility of each positive psychology exercise with a 10-point Likert scale (0=very difficult/not helpful; 10=very easy/very helpful). The mean ease and utility of each exercise and overall will be calculated.
Time Frame: 9 weeks
Population: For the acceptability analysis, the analysis population denominator was 15 participants who received PATH.
Measure: Mean (95% Confidence Interval); unit: score on a 10.0-point scale
Arm/Group | PATH Intervention
Number analyzed (Participants) | 15
score on a 10.0-point scale
  Acceptability - Mean Ease Score | 8.1 [7.4 to 8.7]
  Acceptability - Mean Utility Score | 8.3 [7.8 to 8.9]

ADVERSE EVENTS:
Time Frame: Treatment-related and non-treatment related adverse event data were collected during the active study period, which lasted from study enrollment through follow-up assessment completion (week 9). Because this was a supportive care intervention, adverse events were not assessed at a pre-specified time. Instead, adverse events were recorded as reported by study participants during the active study period.
Description: Treatment-related and non-treatment related adverse event data that were related to study procedures were reported to the Institutional Review Board (IRB) at the PI's discretion. Participants requesting withdrawal from the study were asked to provide reasons for withdrawal to monitor for adverse events or unanticipated events related to study procedures.
Arm/Group | PATH Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT05216978/Prot_SAP_000.pdf